CLINICAL TRIAL: NCT04003792
Title: Treatment With Hepatic Arterial Infusion of Oxaliplatin in Combination With Systemic FOLFIRI Chemotherapy and Bevacuzimab in Patients With Liver-only Colorectal Liver Metastases (CRLM): Conversion to Complete Resection in Patients With Initially Inoperable Liver-only CRLM.
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Eran Sadot, Head of Hepatopancreatobiliary service, Principal Investigator, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 0275-19-RMC
Record Dates: First submitted 2019-06-27; First posted 2019-07-01 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-10

CONDITIONS: Liver Metastasis Colon Cancer
MeSH Terms: interventions — Oxaliplatin; IFL protocol; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- single arm prospective trial (Experimental)
  Interventions: Drug: oxaliplatin; Drug: FOLFIRI Protocol; Drug: Bevacizumab

INTERVENTIONS:
Drug: oxaliplatin — intra-arterial oxaliplatin administration
Drug: FOLFIRI Protocol — systemic FOLFIRI chemotherapy
Drug: Bevacizumab — systemic bevacuzimab therapy

SUMMARY:
A few studies have documented that some patients can be down-staged from an initially inoperable state to a potentially resectable state. Five-year survival in initially inoperable patients that ultimately come to a complete resection appears to be similar to patients who are resected at first presentation. The investigators goal is to assess the rate of conversion to complete resection in patients with initially inoperable liver-only metastases due to colorectal cancer after treatment with HAI of oxaliplatin with FOLFIRI and bevacuzimab systemic treatment.

ELIGIBILITY:
Subject Inclusion Criteria:

* Histologically confirmed colorectal adenocarcinoma metastatic to the liver.
* The patient must have inoperable liver metastases as agreed upon by any two hepatobiliary surgeons and the assigned radiologist.
* A patient may have had prior chemotherapy or be previously untreated.
* ECOG PS <2

Subject Exclusion Criteria:

* Prior radiation, hepatic thermo ablation or resection (other than biopsy) to the liver.
* Patient may not have received prior treatment with hepatic artery infusion (HAI).
* Extrahepatic metastases
* Female patients who are pregnant or lactating

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2022-01 (Estimated); Study Completion 2022-01 (Estimated)

PRIMARY OUTCOMES:
conversion rate to complete resection in patients with initially inoperable liver-only metastases due to colorectal cancer after treatment with HAI of oxaliplatin with FOLFIRI and bevacuzimab systemic treatment. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No